CLINICAL TRIAL: NCT06793475
Title: Aponermin-Based Bridging Therapy Prior to CAR-T Infusion in Relapsed/Refractory Multiple Myeloma Patients With Extramedullary Disease: A Prospective, Single-Arm, Multicenter, Open-Label Study
Brief Title: Aponermin-Based Bridging Therapy Prior to CAR-T Infusion in Relapsed/Refractory Multiple Myeloma Patients With Extramedullary Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024113
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-12

CONDITIONS: Extramedullary Multiple Myeloma
MeSH Terms: interventions — carfilzomib; Thalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aponermin-based regimen bridging CAR-T therapy (Experimental): Patients will receive aponermin-based bridging therapy followed by Fc-based conditioning and CAR-T cell infusion. One month after CAR-T cell therapy, patients will begin maintenance therapy for at most 6 months or until disease progression, death, intolerance, withdrawal for other reasons, or the study's termination/completion.
  Interventions: Biological: anti-BCMA/GPRC5D bispecific CAR-T; Drug: Apornemin; Drug: Carfilzomib; Drug: Thalidomide; Drug: Dexamethasone

INTERVENTIONS:
Biological: anti-BCMA/GPRC5D bispecific CAR-T — Autologous BCMA/GPRC5D bispecific CAR-T cells, infusion intravenously at a target dose of 2-4 x 10^6 anti-BCMA/GPRC5D bispecific CAR-T cells/kg.
Drug: Apornemin — Apornemin 10mg/kg will be administered by i.v. infusion. Apornemin will be administered on Days 1-5, 15-19 during bridging therapy, and on Days 1-5 every 28-day cycle during maintanance treatment.
Drug: Carfilzomib — Carfilzomib 27mg/m^2 will be administered by i.v. on Days 1,2,8,9 during bridging therapy.
Drug: Thalidomide — Thalidomide (150mg/d) will be administered by p.o. on Days 1-14 during bridging therapy, and Days 1-28 every 28-day cycle during maintanance treatment.
Drug: Dexamethasone — Dexamethasone (20mg/d) will be administered by i.v. or p.o. on Days 1-4,8,9 during bridging therapy.

SUMMARY:
This is a prospective, single-arm, multicenter, open-label study to evaluate the efficacy and safety of aponermin-based bridging therapy prior to CAR-T infusion in relapsed/refractory multiple myeloma patients with extramedullary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Be informed and voluntarily sign the Informed Consent Form (ICF).
2. Age ≥18 years.
3. Confirmed diagnosis of Multiple Myeloma(MM) (IMWG consensus guidelines)
4. Subjects with diagnosed relapsed or refractory extramedullary multiple myeloma according to IMWG criteria and have had at least 1 prior lines of therapy. Extramedullary disease (EMD) is defined as soft-tissue plasmacytomas NOT arising from skeletal lesions. The maximum diameter of extramedullary lesions should ≥2cm detected by physical exam and confirmed (when required) by Weight Bearing CT/MRI/PET-CT and/or biopsy.
5. ECOG score is ≤ 2
6. No active infections.
7. Negative for HBV-DNA, HCV-RNA, and HIV.
8. Liver function meeting the following criteria: Total bilirubin <1.5 × ULN (patients with Gilbert's syndrome must have total bilirubin <3 × ULN), ALT and AST <3 × ULN.
9. Renal function meeting the following criteria: Creatinine clearance ≥30mL/min (calculated using the Cockcroft-Gault formula).
10. Blood tests conducted within 7 days before screening must meet the following standards: WBC count ≥1.0×10⁹/L, Hemoglobin ≥70g/L, Platelet count ≥75×10⁹/L or ≥50×10⁹/L (if ≥50% plasma cells are present in bone marrow); Or as determined appropriate by the investigator.
11. Patients receiving hematopoietic growth factors (e.g., erythropoietin, granulocyte colony-stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor [GM-CSF], and platelet-stimulating factors such as thrombopoietin [TPO] or interleukin-11) must stop such treatments at least 2 weeks prior to screening.
12. Non-pregnant female patients must confirm pregnancy negativity at screening (via β-hCG serum test or urine pregnancy test).
13. Male patients, female patients of childbearing potential, and their partners must agree to use effective contraception during the treatment period and for at least 3 months after CAR-T cell infusion.
14. Male patients must agree not to donate sperm, starting from the initial screening period until 90 days after the last dose.
15. Patients must agree to comply with study procedures and follow-up visits.

Exclusion Criteria:

1. Plasma cell leukemia or solitary plasmacytoma.
2. Prior exposure to both BCMA- and GPRC5D-targeted therapies (patients who have received only one of these targeted therapies are eligible for enrollment).
3. Evidence of primary or secondary resistance to elotuzumab, carfilzomib, or thalidomide.
4. Pregnant or breastfeeding women, or women with pregnancy plans within the next six months.
5. Infectious diseases (e.g., HIV, active tuberculosis, etc.).
6. Active hepatitis B or hepatitis C infection.
7. Abnormal vital signs or inability to cooperate with examinations.
8. Mental or psychological disorders preventing compliance with treatment or treatment evaluation.
9. Severe allergic constitution or severe allergic history, particularly to aponermin, carfilzomib, thalidomide, dexamethasone or other effective components or excipients of related drugs.
10. Significant dysfunction of major organs, such as the heart, lungs, or brain.

9) Patients with severe autoimmune diseases. 11) Any other reasons deemed unsuitable for participation in this study as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | within 1 months after BCMA/GPRC5D CAR-T infusion
  The definition of ORR is the proportion of participants who achieve a PR or better as the best response according to the IMWG criteria.

SECONDARY OUTCOMES:
ORR before CAR-T cell infusion | before CAR-T cell infusion
  ORR before CAR-T cell infusion is defined as the proportion of participants who achieve a confirmed PR or better as the best response after conditioning treatment but prior to CAR-T cell infusion.
Progression free survival(PFS) | Up to 2 year
  Progression free survival is defined as the time from the start of Aponermin treatment to disease progression, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to 2 year
  Overall Survival (OS) is defined as the time from the start of Aponermin treatment to the date of the participant's death.
Adverse events and serious adverse events | Up to 2 year
  Adverse events (AEs), serious adverse events (SAEs), and assessments of clinical laboratory values

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gobroad Boren Hospital, Beijing
  - Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin